CLINICAL TRIAL: NCT01539681
Title: Sorafenib Treatment Modalities for HEpatoceLLular Carcinoma Patients in ItAly
Brief Title: Sorafenib in Hepatocellular Carcinoma Clinical Practice in Italy
Acronym: STELLA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16028; NX1110IT (Other: company internal)
Record Dates: First submitted 2011-12-13; First posted 2012-02-27 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Cancer, Liver; Sorafenib; Nexavar
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Subjects should be treated with sorafenib in compliance with the recommendations written in the local product information.However, the decision on the duration and dose of treatment is at the discretion of the prescribing physician.

SUMMARY:
Prospective, non-interventional, multi-center study. Patients affected by Hepatocellular Carcinoma (HCC) who are candidates for systemic therapy and in whom a decision to treat with sorafenib has been made. Aim of this non-interventional, post-marketing study is to evaluate the efficacy of sorafenib in terms of overall survival rate at 12 months in patients with HCC under daily-life treatment conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically/cytologically confirmed HCC or radiographically diagnosed as per AASLD criteria, who are candidates for systemic therapy and for whom a decision to treat with sorafenib has been made
* Patients must have signed the informed consent form
* Patients must have a life expectancy of at least 8 weeks Inclusion criteria must follow the approved local product information.

Exclusion Criteria:

* Prior treatment with sorafenib
* Concomitant participation in other clinical studies Exclusion criteria must follow the approved local product information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatocellular Carcinoma Patients treated in Italy
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Efficacy (analyzed by overall survival rate) of sorafenib under real-life practice conditions in patients with Hepatocellular Carcinoma. | at 1 year

SECONDARY OUTCOMES:
Adverse event collection of sorafenib under real-life practice conditions in patients with Hepatocellular Carcinoma. | every 4 months on average within approx. 2 years
Overall survival | at 1 year
Time to Progression | every 4 months on average within approx. 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Italy